CLINICAL TRIAL: NCT06410703
Title: A Phase Ib/IIa, Dose Escalation, Open-Label Study of Intratumoral CAN1012 Combined With PD-1 in Patients With Unresectable or Metastatic Advanced Solid Tumors
Brief Title: CAN1012 Combined With PD-1 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Canwell Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CW-103
Record Dates: First submitted 2024-05-05; First posted 2024-05-13 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAN1012(0.01mg)+Toripalimab(240mg) (Experimental): CAN1012(0.01mg)+Toripalimab(240mg)
  Interventions: Drug: CAN1012
- CAN1012(0.017mg)+Toripalimab(240mg) (Experimental): CAN1012(0.017mg)+Toripalimab(240mg)
  Interventions: Drug: CAN1012

INTERVENTIONS:
Drug: CAN1012 — CAN1012 IT injection every three weeks (Q3W), Toripalimab will be administered at the approved dose of 240mg IV Q3W
  Other Names: Toripalimab

SUMMARY:
This is a Phase Ia/IIb, open-label, first-in-human, multicenter, single-arm, dose escalation study of intratumoral CAN1012 combined with PD-1 in patients with Unresectable or Metastatic Advanced Solid Tumors who have exhausted options for standard of care therapy.

DETAILED DESCRIPTION:
The scope of the study is to evaluate the safety of the combination therapy of CAN1012 and PD-1 in human, study its efficacy and pharmacokinetics profiles, as well as explore its pharmacodynamic effects and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and willing to comply with the study's requirements.
2. Male or female age ≥ 18 years at screening.
3. Patients with histologically and cytologically confirmed locally advanced or metastatic solid tumors who have been refractory or intolerant to standard therapies or for whom no standard therapy exists.
4. Metastatic or locally advanced solid tumor that has progressed on, is refractory to, or for which there is no efficacious standard of care therapy. Preferred tumor types include the following:

   Carcinoma of skin, melanoma, Merkel cell carcinoma (MCC), breast cancer, head and neck squamous cell carcinoma (HNSCC), sarcoma, cervical carcinoma, and colorectal cancer
5. Performance status of 0-1 on the ECOG Performance Scale.

Exclusion Criteria:

1. Unresolved toxicities from prior therapy, defined as having not resolved to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0) Grade 0 or 1, with exception of endocrinopathies from prior therapy, alopecia, and vitiligo.
2. Treatment with systemic corticosteroids at doses exceeding 10 mg/day prednisone or equivalent.
3. Has an active infection requiring systemic therapy.
4. Unstable/inadequate cardiac function defined as follows:

   1. New York Heart Association Class 3 or 4 congestive heart failure
   2. uncontrolled hypertension
   3. acute coronary syndrome within 6 months
   4. clinical important cardiac arrhythmia
   5. mean corrected QT (QTc) interval corrected for heart rate >450msec（male），>470msec（female）.
5. A history of interstitial lung disease.
6. A history of coagulopathy resulting in uncontrolled bleeding or other bleeding disorders.
7. Participated in a clinical study of an investigational agent within 30 days of screening.
8. Has known psychiatric, substance abuse, or other disorders that would interfere with cooperation with the requirements of the study in the opinion of the investigator.
9. Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 1 year
  Safety and tolerability as determined by assessing dose limiting toxicities, the maximum tolerated dose or maximal assessed dose per protocol in combination with toripalimab (anti-PD-1) with patients.

SECONDARY OUTCOMES:
To determine the MTD and or RP2D of CAN1012 Combined with PD-1 | Monitor a tumor response to the combination therapy according to RECIST 1.1 or iRECIST 1.1 as appropriate.
  Monitor a tumor response to the combination therapy according to RECIST 1.1 or iRECIST 1.1 as appropriate.
To determine the Pharmacokinetics of CAN1012 Combined with PD-1 | 1 year
  Determine CAN1012 concentrations in plasma after IT administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China